CLINICAL TRIAL: NCT02199379
Title: A Phase 1, Open-Label, Single-Dose, Pharmacokinetic and Safety Study of E7080 (24 mg) Administered to Subjects With Mild, Moderate, and Severe Renal Impairment and to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-005
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-01

CONDITIONS: Renal Impairment; Disease Severity
Keywords: renal impairment; disease severity
MeSH Terms: conditions — Renal Insufficiency | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib (Experimental): Lenvatinib will be taken as a single dose of 24 mg consisting of 2 x 10 mg and 1 x 4 mg capsules. Treatment will be administered orally with 240 mL of water following a 10-hour overnight fast.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be taken as a single dose of 24 mg consisting of 2 x 10 mg and 1 x 4 mg capsules. Treatment will be administered orally with 240 mL of water following a 10-hour overnight fast.
  Other Names: E7080

SUMMARY:
The purpose of this multicenter, open-label, non-randomized, single, oral dose, sequential-cohort study was to determine pharmacokinetics and safety of lenvatinib (24 mg) administered to healthy subjects and to subjects with renal impairment.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, single-dose, sequential-cohort trial in subjects with renal impairment and healthy subjects. The study consists of two phases: A Pretreatment Phase and a Treatment Phase. The two periods in the Pretreatment Phase are: (1) the Screening Period (lasting up to 29 days), and (2) the Baseline Period (one day). The Treatment Period of the Treatment Phase lasts 8 days. The study will enroll a sufficient number of subjects so that 24 to 26 subjects complete the study. This will include six subjects with mild renal impairment (Group 1), six subjects with moderate renal impairment (Group 2), four to six subjects with severe renal impairment (Group 3) and eight subjects with normal renal function (Group 4). Subjects determined to be eligible for the protocol will receive a single 24-mg oral dose of E7080 on Day 1. Subjects will be discharged from clinical site on Day 8.

ELIGIBILITY:
Inclusion Criteria

All subjects should meet all of the following criteria to be included in this study:

1. Male or female subjects, ages 18 to 79, inclusive, at the time of informed consent
2. BMI, 18 to 40 kg/m2, inclusive, at Screening
3. Nonsmokers and smokers who smoke no more than 10 cigarettes per day
4. All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [B-hCG] at the Screening Visit or within 72 hours before the first dose of study drug). Females of child-bearing potential, if not practicing total abstinence or having a vasectomised partner with confirmed azoospermia, must agree to use two highly effective methods of contraception: e.g., 1) an intrauterine device (IUD) or intrauterine system (IUS); 2) a barrier method such as a condom or occlusive cup (diaphragm or cervical/vault caps) plus spermicide (foam, gel, cream, etc.); 3) oral, injected, or implanted hormonal contraceptives throughout the entire study period and for 30 days after study drug discontinuation. Use of a double-barrier method (i.e., use at the same time of a condom plus occlusive cup [diaphragm or cervical/vault caps] plus spermicide [foam, gel, cream, etc.]) is accepted as two highly effective methods of contraception. The only subjects who will be exempt from this requirement are postmenopausal women (defined as women who have been amenorrheic for at least 12 consecutive months, in the appropriate age group, without other known or suspected primary cause) or subjects who have been sterilized surgically or who are otherwise proven sterile (i.e., bilateral tubal ligation with surgery at least 1 month prior to dosing, total hysterectomy, or bilateral oophorectomy with surgery at least 1 month prior to dosing). All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
5. Male subjects who are partners of women of childbearing potential must use a condom plus spermicide and their female partners if of childbearing potential must use a highly effective method of contraception (see methods described in Inclusion Criterion No. 4) beginning at least one menstrual cycle prior to starting study drug, throughout the entire study period, and for 30 days after the last dose of study drug, unless the male subjects are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile (see Inclusion Criterion No.4).
6. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

For healthy subjects with normal renal function the following key inclusion criterion will also apply:

1. Creatinine clearance greater than or equal to 90 mL/min.

For subjects with renal impairment, the following key inclusion criteria will also apply:

1. Subjects must have a diagnosis of renal impairment that has been stable, without any change in disease status, for 60 days prior to study screening, as determined by the investigator.
2. Mild (creatinine clearance, 60-89 mL/min), moderate (creatinine clearance, 30-59 mL/min), or severe (creatinine clearance, 15-29 mL/min) renal impairment
3. Other than renal impairment, subjects must have no history of clinically relevant disease or condition (e.g., significant cardiac or hepatic dysfunction, diseases of the gastrointestinal tract or conditions which may impact drug absorption), as determined by the investigator.
4. Subjects with a history of Type I or Type II diabetes are permissible, providing that, in the opinion of the investigator, they have stable disease. Subjects receiving insulin therapy are permissible provided that they have been on a stable treatment for at least 2 weeks prior to study enrollment and continuing through the study.
5. QT interval corrected for heart rate (QTc) calculated by Fridericia's formula (QTcF) interval lesser than or equal to 500 msec at Screening and Baseline.
6. Subjects may be enrolled with joint approval of the principal investigator (PI) and medical monitor based on subject history and stability of the renal impairment.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

All Subjects:

1. Use of any new medication, including multivitamins, or investigational drug within 14 days prior to the drug administration, or within five times the elimination half-life, whichever is longest, except combined oral contraceptives and occasional use of paracetamol or ibuprofen within 14 days and any local anesthetic within 3 days before study drug administration. Current over-the-counter (OTC) drugs and prescription medication use is permitted, but must be stable and consistent for at least 14 days prior to Screening and throughout the study treatment period.
2. Positive HIV screening test
3. Presence of acute, active liver disease or acute liver injury as indicated by (1) an abnormal liver function test, or (2) clinical or laboratory signs of acute, active hepatitis A, B, or C
4. Systolic blood pressure greater than or equal to 160 mm Hg and/or diastolic blood pressure greater than or equal to 100 mm Hg for healthy subjects and subjects with mild renal impairment; systolic blood pressure greater than or equal to 180 mm Hg and/or diastolic blood pressure greater than or equal to 110 mm Hg for subjects with moderate and severe renal impairment. Readings are to be confirmed by repeat determinations one hour after the first measurement.

Healthy Subjects:

In addition to the Key Exclusion Criteria above for all subjects, other standard exclusion criteria for healthy subjects in Phase 1 studies will be used. These include:

1. Subjects who had a clinically significant illness which required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
2. Subjects with a history of myocardial infarction or active ischemic heart disease
3. Subjects with a disease that may influence the outcome of the study, such as psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism within 4 weeks prior to dosing
4. Gastrointestinal malabsorption or any other condition that may affect PK profiles of E7080 including a history of gastrointestinal surgery (hepatectomy, digestive organ resection, etc.) (Appendectomy and cholecystectomy are, however, permitted.)
5. Subjects with a history of clinically significant drug or food allergies or presently experiencing significant seasonal allergies
6. Subjects who experienced a weight loss or gain of greater than 10% between Screening and prior to dosing
7. Subjects with a QTc interval greater than 450 msec demonstrated on repeated electrocardiogram (ECG) at Screening
8. Subjects with hemoglobin level less than 12.0 g/dL
9. Significant findings revealed by the history, physical or clinical laboratory testing
10. Subjects with a known or suspected history of drug or alcohol misuse within 6 months prior to Screening, or who have a positive urine drug or alcohol test at Screening or Baseline
11. Subjects who have consumed caffeinated beverages or food within 72 hours prior to dosing
12. Receipt of another investigational drug or device within 4 weeks prior to dosing or five half-lives of the other investigational drug, whichever is longer
13. Subjects who received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within one week of dosing
14. Subjects who have engaged in heavy exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters, etc.)
15. Subjects who are unwilling to abide by the requirements of the study, or in the opinion of the investigator, are not likely to complete the study.

Subjects with Renal Impairment:

1. A history of renal transplant
2. Known significant bleeding diathesis (e.g., history of recent bleeding from esophageal varices), which could preclude multiple venipuncture or deep intramuscular injection
3. Significant acute, new onset illness within 2 weeks prior to study drug administration. In addition to the Key Exclusion Criteria above for All Subjects and for Subjects with Renal Impairment, other standard exclusion criteria for healthy subjects in Phase 1 studies will be used for subjects with renal impairment. These include:
4. Subjects who had a clinically significant illness, where said illness is unrelated to their renal impairment, which required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
5. Subjects with a history of significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II; unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment
6. Subjects with a disease that may influence the outcome of the study, such as psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism within 4 weeks prior to dosing
7. Gastrointestinal malabsorption or any other condition that may affect PK profiles of E7080 including a history of gastrointestinal surgery (hepatectomy, digestive organ resection, etc.). (Appendectomy and cholecystectomy are, however, permitted.)
8. Subjects with a known history of clinically significant drug or food allergies or presently experiencing significant seasonal allergies
9. Subjects who experienced a weight loss or gain of greater than 10% between Screening and prior to dosing
10. Significant findings revealed by the history, physical or clinical laboratory testing where said findings are unrelated to the subject's renal impairment
11. Subjects with a known or suspected history of drug or alcohol misuse within 6 months prior to Screening, or who have a positive urine drug or alcohol test at Screening or Baseline
12. Subjects who have consumed caffeinated beverages or food within 72 hours prior to dosing
13. Receipt of another investigational drug or device within 4 weeks prior to dosing or five half-lives of the other investigational drug, whichever is longer
14. Subjects who received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within one week of dosing
15. Subjects who have engaged in heavy exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters, etc.)
16. Subjects who are unwilling to abide by the requirements of the study, or in the opinion of the investigator, are not likely to complete the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of lenvatinib: Cmax | Day 1 to Day 8
Pharmacokinetics of lenvatinib: AUC(0-inf) | Day 1 to Day 8
Pharmacokinetics of lenvatinib: AUC(0-t) | Day 1 to Day 8

SECONDARY OUTCOMES:
Safety as Measured by Outcome of all Adverse Events (AEs) | Screening, Baseline and Treatment period (Day 1 to Day 8)
Safety as Measured by Outcome of treatment-emergent AEs (TEAEs) | Screening, Baseline and Treatment period (Day 1 to Day 8)
Safety as Measured by Outcome of serious adverse events (SAEs) | Screening, Baseline and Treatment period (Day 1 to Day 8)
Safety as Measured by Laboratory Values | Screening, Baseline and Treatment period (Day 1 to Day 8)
Safety as Measured by vital signs | Screening, Baseline and Treatment period (Day 1 to Day 8)
Safety as Measured by ECGs | Screening, Baseline and Treatment period (Day 1 to Day 8)
Safety as Measured by performance of physical examinations. | Screening, Baseline and Treatment period (Day 1 to Day 8)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Knoxville, Tennessee